CLINICAL TRIAL: NCT01193296
Title: Prospective, Randomized, Open-label Study With Blinded Endpoint (PROBE Design) to Compare the 72 hr Glycemic Profiles Obtained by Continuous Subcutaneous Glucose Monitoring (CSGM) in Type 2 Diabetic Patients at Baseline With Metformin Monotherapy and After an 8-week Period With the Addition of Either Vildagliptin or Sitagliptin in Patients Insufficiently Controlled by Metformin After at Least 3 Months of Monotherapy
Brief Title: Glycemic Holter Study (Continuous Glucose Monitoring) -
Acronym: OPTIMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AFR02
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus, vildagliptin, continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vildagliptin; Sitagliptin Phosphate

ARMS (2):
- Vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Vildagliptin
  Arms: Vildagliptin
Drug: Sitagliptin
  Arms: Sitagliptin

SUMMARY:
The study will assess glycemic variability and optimized glycemic control in T2DM patients treated with a DPP-4 inhibitor as add-on therapy to metformin.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus (DM) willing to perform SMBG at least 6 times daily to use the MiniMed CGMS for up to 3 consecutive days on 2 occasions.
* HbA1c: 6.5 to 9% with metformin monotherapy for a least 3 months

Exclusion Criteria:

* Age >= 80 years
* BMI <= 22 and >=40 kg/m2
* Secondary T2 DM
* Hepatic failure, ASAT/ALAT>3 ULN, and moderate/severe renal failure (CI < 50 ml/min) CHF III & IV

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Glycemic variability assessed by MAGE (Mean Amplitude of Glycemic Excursion) | 8 weeks

SECONDARY OUTCOMES:
Glycemic control assessed through CSGM | 8 weeks
Glycemic control assessed by A1C, FPG, PPG and the mean of 6 points self-monitoring of blood glucose (SMBG) at baseline and after 8 weeks | 8 weeks
Unrecognized hypoglycemic periods recorded by CSGM, frequency and duration | 8 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Investigative Site, Bondy
  - Investigative Site, Corbeil
  - Investigative Site, Marseille
  - Investigative Site, Nancy
  - Investigative Site, Paris
  - Investigative Site, Toulouse
  - Investigative Site, Vénissieux

REFERENCES:
- [Derived] Guerci B, Monnier L, Serusclat P, Petit C, Valensi P, Huet D, Raccah D, Colette C, Quere S, Dejager S. Continuous glucose profiles with vildagliptin versus sitagliptin in add-on to metformin: results from the randomized Optima study. Diabetes Metab. 2012 Oct;38(4):359-66. doi: 10.1016/j.diabet.2012.06.001. Epub 2012 Jul 17. PMID 22809630
- [Derived] Monnier L, Colette C, Comenducci A, Vallee D, Dejager S. Add-on therapies to metformin in type 2 diabetes: what modulates the respective decrements in postprandial and basal glucose? Diabetes Technol Ther. 2012 Oct;14(10):943-50. doi: 10.1089/dia.2012.0045. Epub 2012 Jul 9. PMID 22775317